CLINICAL TRIAL: NCT05458297
Title: A Multicenter, Open-label, Phase 2 Basket Study to Evaluate the Safety and Efficacy of MK-2140 as a Monotherapy and in Combination in Participants With Aggressive and Indolent B-cell Malignancies (waveLINE-006)
Brief Title: A Study of Zilovertamab Vedotin (MK-2140) as Monotherapy and in Combination in Participants With Aggressive and Indolent B-cell Malignancies (MK-2140-006)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2140-006; MK-2140-006 (Other: MSD); jRCT2011230019 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2022-501374-19-00 (Registry Identifier: EU CT); U1111-1280-1849 (Registry Identifier: UTN); 2021-004450-36 (EudraCT Number)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Follicular Lymphoma; Richter Transformation Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A, Relapsed or Refractory MCL with 2 Prior Lines of Therapy (Experimental): Participants will receive zilovertamab vedotin intravenous (IV) infusion at Dose 1 every 3 weeks (Q3W) until disease progression or discontinuation.
  Interventions: Biological: Zilovertamab vedotin
- Cohort B, Relapsed or Refractory RT with 1 Prior Line of Therapy (Experimental): Participants will receive zilovertamab vedotin IV infusion at Dose 1 every 3 weeks (Q3W) until disease progression or discontinuation.
  Interventions: Biological: Zilovertamab vedotin
- Cohort C, Relapsed or Refractory MCL with 1 Prior Line of Therapy (Experimental): Participants will receive zilovertamab vedotin IV infusion at Dose 2 every 3 weeks (Q3W) combined with nemtabrutinib oral dose daily until disease progression or discontinuation.
  Interventions: Biological: Zilovertamab vedotin; Drug: Nemtabrutinib
- Cohort D, Relapsed or Refractory FL and CLL with 2 Prior Lines of Therapy (Experimental): Participants will receive either zilovertamab vedotin IV infusion Dose 1 every 3 weeks (Q3W) until disease progression or discontinuation.
  Interventions: Biological: Zilovertamab vedotin
- Cohort E, Relapsed or Refractory FL with 2 Prior Lines of Therapy (Experimental): Participants will receive either zilovertamab vedotin IV infuison Dose 1 every 3 weeks (Q3W) until disease progression or discontinuation.
  Interventions: Biological: Zilovertamab vedotin

INTERVENTIONS:
Biological: Zilovertamab vedotin — IV infusion
  Other Names: MK-2140
Drug: Nemtabrutinib — Oral tablet
  Other Names: MK-1026
  Arms: Cohort C, Relapsed or Refractory MCL with 1 Prior Line of Therapy

SUMMARY:
The purpose of this study is to assess the safety and tolerability of zilovertamab vedotin as monotherapy and in combination in participants with select B-cell lymphomas including mantle cell lymphoma (MCL), Richter's transformation lymphoma (RTL), follicular lymphoma (FL), and chronic lymphocytic leukemia (CLL). This study will also evaluate zilovertamab vedotin as monotherapy and in combination with respect to objective response rate.

* Cohort A: Participants with relapsed or refractory MCL relapsed or refractory disease after at least 2 prior systemic therapies including a Bruton's tyrosine kinase inhibition/inhibitor (BTKi), and post therapy chimeric antigen receptor T (CAR-T) cell therapy or ineligible for CAR-T cell therapy
* Cohort B: Participants with relapsed or refractory RT disease after at least 1 prior systemic therapy
* Cohort C: Participants with relapsed or refractory MCL relapsed or refractory disease after at least 1 prior systemic therapy and no prior exposure to a non-covalent BTKi
* Cohort D: Participants with relapsed or refractory FL and CLL relapsed or refractory disease after at least 2 prior systemic therapies and have no other available therapy
* Cohort E: Participants with relapsed or refractory FL after at least 2 prior systemic therapies and have no other available therapy

The primary study hypothesis is that zilovertamab vedotin monotherapy has an increased Objective Response Rate (ORR) per Lugano Response Criteria as assessed by blinded independent central review (BICR).

As of Amendment 07, Cohort D is closed to enrollment of participants with CLL and enrollment of participants into Arm 2 (zilovertamab vedotin at Dose 2 on Days 1 & 8 of each 3 Week Cycle (Q2/3W)).

ELIGIBILITY:
The main inclusion criteria include, but are not limited to the following:

Inclusion Criteria:

* For aggressive B-cell malignancies mantle cell lymphoma (MCL): Has histologically confirmed biopsy according to the 2016 World Health Organization (WHO) classification of neoplasms of the hematopoietic and lymphoid tissues and has relapsed or refractory disease after at least 2 prior systemic therapies including a Bruton's tyrosine kinase inhibition/inhibitor(s) (BTKi), and is post chimeric antigen receptor T (CAR-T) cell therapy or is ineligible for CAR-T cell therapy.
* For aggressive B-cell malignancies MCL Cohort C: Has histologically confirmed biopsy according to the 2016 World Health Organization (WHO) classification of neoplasms of the hematopoietic and lymphoid tissues and has relapsed or refractory disease after at least 1 prior systemic therapy and has no prior exposure to a non-covalent BTKi.
* For aggressive B-cell malignancies Richter transformation lymphoma (RTL): Has histologically confirmed biopsy according to the 2016 World Health Organization (WHO) classification of neoplasms of the hematopoietic and lymphoid tissues and has relapsed or refractory disease.
* For indolent B-cell malignancies follicular lymphoma (FL) and chronic lymphocytic leukemia (CLL): Has histologically confirmed biopsy and has relapsed or refractory disease after at least 2 prior systemic therapies and no other available therapy.
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization/allocation.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 assessed within 7 days before cycle 1 day 1.

Exclusion Criteria:

* Has received solid organ transplant at any time.
* Has clinically significant (ie, active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina (<6 months prior to enrollment), congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication.
* Has pericardial effusion or clinically significant pleural effusion.
* Has ongoing Grade >1 peripheral neuropathy.
* Has a demyelinating form of Charcot-Marie-Tooth disease.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
* Participants with FL who have transformed to a more aggressive type of lymphoma.
* Has received prior systemic anticancer therapy within 5 half-lives or 4 weeks (if prior therapy was a monoclonal antibodies) or 2 weeks (if prior therapy was small molecules like kinase inhibitors) prior to the first dose of study intervention.
* Has received prior radiotherapy within 28 days of start of study intervention. Participants must have recovered from all radiation-related toxicities.
* Has ongoing corticosteroid therapy exceeding 30 mg daily of prednisone equivalent.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Has known active central nervous system (CNS) lymphoma involvement or active CNS involvement by lymphoma.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection not well controlled on antiretroviral therapy (ART)
* Active HBV or hepatitis C virus (HCV) infection.
* For Cohort C only: has any clinically significant gastrointestinal abnormalities that might alter absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2029-05-17 (Estimated); Study Completion 2029-05-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with MCL (Cohort C), FL (Cohort D), and CLL with ≥1 Adverse Event (AE) | Up to approximately 81 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with MCL (Cohort C), FL (Cohort D), and CLL who experienced an AE will be reported.
Percentage of Participants with MCL (Cohort C), FL (Cohort D), and CLL who Discontinue from Study Therapy Due to AE | Up to approximately 81 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with MCL (Cohort C), FL (Cohort D), and CLL who discontinued study treatment due to an AE will be reported.
Percentage of Participants with MCL (Cohort C) who Experience a Dose-Limiting Toxicity (DLT) | Up to approximately 81 months
  The Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 will be used to grade the severity of AEs. DLTs for participants with MCL (Cohort C) as assessed by investigator will be reported.
Objective Response Rate (ORR) per Lugano Response Criteria as Assessed by Blinded Independent Central Review (BICR) in Participants with MCL (Cohort A), RT, and FL (Cohorts D & E) | Up to approximately 81 months
  ORR, defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per Lugano Response Criteria as assessed by BICR in Participants with MCL (Cohort A), RT, and FL (Cohorts D & E) will be reported.
ORR per Lugano Response Criteria as Assessed by Investigator in Participants with MCL (Cohort C) | Up to approximately 81 months
  ORR, defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per Lugano Response Criteria as assessed by investigator in Participants with MCL (Cohort C) will be reported.
ORR per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria as Assessed by Investigator in Participants with CLL | Up to approximately 81 months
  ORR, defined as the percentage of participants who achieve a CR or PR per iwCLL criteria as assessed by investigator in participants with CLL will be reported.

SECONDARY OUTCOMES:
Duration of Response (DOR) per Lugano Response Criteria as Assessed by BICR in Participants with MCL (Cohort A), RT, and FL (Cohorts D & E) | Up to approximately 81 months
  DOR, defined as the time from the first documented evidence of CR or PR per Lugano Response Criteria as assessed by BICR, until disease progression or death due to any cause, whichever occurs first, in Participants with MCL (Cohort A), RT, and FL (Cohorts D & E) will be reported.
DOR per Lugano Response Criteria as Assessed by Investigator in Participants with MCL (Cohort C) | Up to approximately 81 months
  DOR, defined as the time from the first documented evidence of CR or PR per Lugano Response Criteria as assessed by investigator, until disease progression or death due to any cause, whichever occurs first, in participants with MCL (Cohort C) will be reported.
DOR per iwCLL Criteria as Assessed by Investigator in Participants with CLL | Up to approximately 81 months
  DOR, defined as the time from the first documented evidence of CR or PR per iwCLL criteria as assessed by investigator, until disease progression or death due to any cause, whichever occurs first, in participants with CLL will be reported.
Percentage of Participants with ≥1 AE in Participants with MCL (Cohort A), RT, and FL (Cohort E) | Up to approximately 81 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with MCL (Cohort A), RTL, and FL (Cohort E) who experienced an AE will be reported.
Percentage of Participants Discontinuing from Study Therapy Due to AE in Participants with MCL (Cohort A), RT, and FL (Cohort E) | Up to approximately 81 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with MCL (Cohort A), RT, and FL (Cohort E) who discontinued study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (109):
- United States (20):
  - Alaska Oncology and Hematology ( Site 0037), Anchorage, Alaska
  - Banner MD Anderson Cancer Center ( Site 0040), Gilbert, Arizona
  - Banner MD Anderson Cancer Center - University Medical Center Phoenix-Medical Oncology ( Site 0036), Phoenix, Arizona
  - University of Colorado Anschutz Medical Campus-The Center for Cancer and Blood Disorders ( Site 0008), Aurora, Colorado
  - Cancer Care Specialists of Illinois ( Site 0031), Decatur, Illinois
  - University of Kansas Medical Center-Division of Hematologic Malignancies and Cellular Therapeutics ( Site 0038), Fairway, Kansas
  - Norton Women's and Children's Hospital-Norton Cancer Institute - St. Matthews ( Site 0007), Saint Matthews, Kentucky
  - Greenebaum Comprehensive Cancer Center-Hematology & Multiple Myeloma ( Site 0010), Baltimore, Maryland
  - Tufts Medical Center ( Site 0024), Boston, Massachusetts
  - Massachusetts General Hospital ( Site 0018), Boston, Massachusetts
  - Dana-Farber Cancer Institute-Lymphoma ( Site 0026), Boston, Massachusetts
  - University of Michigan ( Site 0009), Ann Arbor, Michigan
  - Henry Ford Hospital ( Site 0035), Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai ( Site 0023), New York, New York
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0014), Fargo, North Dakota
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C ( Site 0004), Columbus, Ohio
  - Avera Cancer Institute- Research ( Site 0011), Sioux Falls, South Dakota
  - Medical Oncology Associates, PS ( Site 0005), Spokane, Washington
  - University of Wisconsin Hospitals and Clinics-Carbone Cancer Center ( Site 0030), Madison, Wisconsin
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0021), Milwaukee, Wisconsin
- Brazil (4):
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 1807), Natal, Rio Grande do Norte
  - Instituto Nacional de Câncer - INCA-Divisão de Pesquisa Clínica e Desenvolvimento Tecnológico HC1 ( Site 1809), Rio de Janeiro
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 1808), São Paulo
  - Hospital Paulistano-Americas Oncologia ( Site 1805), São Paulo
- Canada (7):
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 0201), Vancouver, British Columbia
  - The Moncton Hospital-Oncology ( Site 0211), Moncton, New Brunswick
  - QEII Health Sciences Centre - Victoria General Site ( Site 0213), Halifax, Nova Scotia
  - London Health Sciences Centre ( Site 0203), London, Ontario
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0200), Toronto, Ontario
  - Jewish General Hospital ( Site 0202), Montreal, Quebec
  - Allan Blair Cancer Centre-Care Services ( Site 0208), Regina, Saskatchewan
- Chile (4):
  - IC La Serena Research ( Site 1909), La Serena, Coquimbo Region
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 1907), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 1910), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago ( Site 1903), Santiago, Region M. de Santiago
- China (16):
  - Beijing Cancer hospital ( Site 1200), Beijing, Beijing Municipality
  - Zhujiang Hospital ( Site 1207), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 1202), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center ( Site 1201), Guangzhou, Guangdong
  - Henan Cancer Hospital-hematology department ( Site 1212), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 1210), Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 1221), Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University-hematology department ( Site 1218), Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 1223), Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 1204), Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital ( Site 1213), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital-oncology department ( Site 1220), Chuangchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 1208), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University-Head and Neck Oncology ( Site 1206), Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University ( Site 1211), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 1214), Hangzhou, Zhejiang
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice-Interni hematologicka a onkologicka klinika ( Site 0300), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Klinika Hematoonkologie ( Site 0301), Ostrava, Moravskoslezský kraj
  - Vseobecna fakultni nemocnice v Praze-I. Interní klinika - klinika hematologie ( Site 0302), Prague
- North Estonia Medical Centre Foundation ( Site 0401), Tallinn, Harju, Estonia
- Germany (2):
  - Universitaetsklinikum Ulm. ( Site 0502), Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Koeln ( Site 0506), Cologne, North Rhine-Westphalia
- St. James's Hospital ( Site 0600), Dublin, Ireland
- Israel (7):
  - Emek Medical Center-Hematology Unit ( Site 0705), Afula
  - Soroka Medical Center-Hematology Department ( Site 0707), Beersheba
  - Rambam Health Care Campus-Hematology and Bone Marrow Transplantation ( Site 0706), Haifa
  - Carmel Hospital ( Site 0709), Haifa
  - Hadassah Medical Center ( Site 0701), Jerusalem
  - Galilee Medical Center ( Site 0710), Nahariya
  - Sheba Medical Center-Hemato Oncology ( Site 0700), Ramat Gan
- Italy (4):
  - IRCCS - AOU di Bologna-SSD: Diagnosi e terapie dei linfomi e delle sindromi linfoproliferative cron ( Site 0800), Bologna, Emilia-Romagna
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 0802), Rozzano, Milano
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare -Azienda Ospedaliera Nazionale SS. Ant ( Site 0803), Alessandria
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -ISTITUTO DI EMATOLOGIA ( Site 0804), Roma
- Japan (9):
  - National Hospital Organization Nagoya Medical Center ( Site 1108), Nagoya, Aichi-ken
  - Hokkaido University Hospital ( Site 1104), Sapporo, Hokkaido
  - Tokai University Hospital ( Site 1100), Isehara, Kanagawa
  - Tohoku University Hospital ( Site 1106), Sendai, Miyagi
  - Kindai University Hospital ( Site 1102), Sakai, Osaka
  - National Cancer Center Hospital ( Site 1103), Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 1101), Koto, Tokyo
  - Kyushu University Hospital ( Site 1105), Fukuoka
  - Okayama University Hospital ( Site 1107), Okayama
- Peru (2):
  - Centro Medico Monte Carmelo ( Site 1702), Arequipa, Ariqipa
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS ( Site 1700), Lima
- Poland (6):
  - Pratia MCM Krakow ( Site 1001), Krakow, Lesser Poland Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej-Oddzial Hematologiczny ( Site 1006), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Chłonnego ( Site 1002), Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej MSWiA w Olsztynie-Oddzial Kliniczny Hematologii ( Site 1007), Olsztyn, Warmian-Masurian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumat-Oddiał Hematologii Ogólnej ( Site 1008), Lodz, Łódź Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Hematologii i Transplantacji S ( Site 1010), Kielce, Świętokrzyskie Voivodeship
- Portugal (3):
  - Champalimaud Foundation ( Site 2002), Lisbon, Lisbon District
  - Unidade Local de Saude de Braga - Hospital de Braga ( Site 2001), Braga
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 2000), Porto
- National Cancer Centre Singapore ( Site 1500), Singapore, Central Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital ( Site 1300), Seoul
  - Samsung Medical Center ( Site 1301), Seoul
- Spain (5):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Haematology Department ( Site 4003), L'Hospitalet Del Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 4004), Barcelona, Catalonia
  - MD Anderson Cancer Center ( Site 4006), Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra ( Site 4005), Pamplona, Navarre
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca-Hematology ( Site 4001), Salamanca
- Sweden (3):
  - Skånes Universitetssjukhus Lund ( Site 5000), Lund, Skåne County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 5002), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset ( Site 5003), Gothenburg, Västra Götaland County
- Turkey (Türkiye) (5):
  - Mega Medipol-Hematology ( Site 6009), Stanbul, Istanbul
  - Ege Universitesi Hastanesi ( Site 6002), Bornova, İzmir
  - Ankara Universitesi Tip Fakultesi Hastanesi-hematology ( Site 6001), Ankara
  - Trakya University ( Site 6005), Edirne
  - Ondokuz Mayıs Universitesi-Oncology department ( Site 6004), Samsun
- United Kingdom (4):
  - The Royal Cornwall Hospital-Haematology ( Site 7006), Truro, Cornwall
  - University College London Hospital ( Site 7001), London, London, City of
  - The Churchill Hospital ( Site 7002), Oxford, Oxfordshire
  - The Christie NHS Foundation Trust ( Site 7007), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26306&tenant=MT_MSD_9011